CLINICAL TRIAL: NCT06917963
Title: Study of Treatment With Intensified Omeprazole Treatment to Prevent High Output Stoma 1: a Randomized, Non-blinded, Controlled Trial
Brief Title: Study of Treatment With Intensified Omeprazole Treatment to Prevent High Output Stoma 1
Acronym: STOP-HOS-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Tomasz Sylwestrzak, Medical Doctor, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB/99/2025
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Stoma - Ileostomy; High Output Stoma; Colon Cancer; IBD (Inflammatory Bowel Disease); Ileus; Omeprazole
Keywords: stoma; ileostomy; high output stoma; omeprazole; ipp; colon cancer; ibd
MeSH Terms: conditions — Colonic Neoplasms; Inflammatory Bowel Diseases; Ileus; Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensified Treatment Arm (Experimental): Participants in this group will receive intensified therapy, starting with an initial intravenous loading dose of 80 mg of omeprazole, followed by 40 mg administered intravenously twice daily (morning and evening) during hospitalization and after discharge to complete 10 days of omeprazole therapy.
  Interventions: Drug: Intensified intravenous omeprazole therapy (loading dose 80 mg IV, then 40 mg IV twice daily at 6:00 AM and 6:00 PM)
- Standard Treatment Arm (Active Comparator): Participants in this group will receive the standard therapy consisting of a single daily intravenous dose of omeprazole (40 mg), administered each morning during hospitalization.
  Interventions: Drug: Standard intravenous omeprazole therapy (40 mg IV once daily at 6:00 AM).

INTERVENTIONS:
Drug: Intensified intravenous omeprazole therapy (loading dose 80 mg IV, then 40 mg IV twice daily at 6:00 AM and 6:00 PM) — This intervention consists of intensified intravenous omeprazole therapy specifically designed to reduce high-output ileostomy after surgery. It includes an initial loading dose of 80 mg omeprazole administered intravenously on the day before surgery (or on the day of surgery in emergency cases), followed by a continuous treatment of 40 mg intravenously twice daily (at 6:00 AM and 6:00 PM) during hospitalization and after discharge to complete 10 day therapy, distinguishing it from standard once-daily omeprazole dosing protocols typically used for gastrointestinal ulcer prophylaxis.
  Arms: Intensified Treatment Arm
Drug: Standard intravenous omeprazole therapy (40 mg IV once daily at 6:00 AM). — The control group will receive standard intravenous omeprazole therapy as per routine clinical practice for gastrointestinal prophylaxis. Participants will receive a single daily dose of 40 mg omeprazole intravenously administered at 6:00 AM during hospitalization. This standard dosing regimen serves as the comparator for assessing the efficacy of the intensified dosing regimen used in the experimental group.
  Arms: Standard Treatment Arm

SUMMARY:
The goal of this clinical trial is to evaluate if intensified omeprazole therapy can reduce high-output stoma (HOS) in adults undergoing ileostomy formation surgery. The main objectives of the study are:

* To assess if intensified omeprazole treatment significantly reduces mean daily ileostomy output (ml/24h) during the first three postoperative days compared to standard omeprazole treatment.
* To evaluate the proportion of patients meeting the criteria for high-output stoma (HOS ≥1400 ml/day) on consecutive postoperative days.
* To measure the time required for stabilization of ileostomy output (<1400 ml/day maintained for three consecutive days).
* To determine the incidence of dehydration-related complications, specifically electrolyte disturbances (hyponatremia, hypokalemia).
* To compare the length of initial hospital stay, frequency of rehospitalizations within 30 days post-discharge, and total length of hospital stay (including rehospitalizations).

Researchers will compare 10 days intensified omeprazole treatment (loading dose of 80 mg IV followed by 40 mg IV twice daily) with standard treatment (40 mg IV once daily) to determine the effectiveness of intensified dosing in reducing ileostomy output and improving postoperative outcomes.

Participants will:

* Receive either standard or intensified intravenous omeprazole during their hospitalization and after discharge for 10 days combined.
* Undergo daily measurements of ileostomy output.
* Have routine laboratory assessments of electrolyte levels.
* Participate in follow-up assessments up to 30 days post-discharge, conducted either through outpatient visits or telephone consultations.

DETAILED DESCRIPTION:
This clinical trial investigates whether intensified omeprazole therapy can effectively reduce a condition known as high-output stoma (HOS) in adult patients undergoing ileostomy surgery. Ileostomy surgery involves creating an opening in the abdomen (stoma) to divert waste away from a diseased or surgically removed section of the intestine. After this procedure, some patients develop an excessive fluid output from the stoma, known as high-output stoma, defined as the production of more than 1400 ml of fluid per day. This excessive fluid loss can cause serious health issues, including severe dehydration, electrolyte imbalances (such as low sodium or potassium levels), nutritional deficiencies, increased risk of kidney problems, cardiovascular complications, and prolonged hospital stays.

Currently, the standard treatment for managing high-output stoma includes dietary changes, restricting fluid intake, administering anti-diarrheal medications like loperamide, and providing intravenous fluids and electrolytes. However, many patients continue to experience high stoma output despite these standard treatments.

Previous studies have suggested that proton pump inhibitors (PPIs) such as omeprazole, medications commonly used to reduce stomach acid, may help decrease the total amount of intestinal fluid produced. Omeprazole increases the pH level (reduces acidity) of the stomach contents, which might reduce irritation in the intestine and slow down fluid loss from the stoma. Although initial results are promising, current data are limited.

In this randomized clinical trial, researchers aim to determine if providing an intensified dosing regimen of omeprazole can significantly reduce ileostomy fluid output and improve clinical outcomes compared to the standard dosing. The study will include adult patients scheduled for elective or emergency ileostomy surgery.

Participants will be randomly assigned to one of two groups:

* Standard treatment group: Participants will receive the standard hospital treatment, which includes a daily intravenous dose of 40 mg omeprazole each morning.
* Intensified treatment group: Participants will receive an intensified regimen of omeprazole, starting with an initial intravenous loading dose of 80 mg, followed by 40 mg given twice daily (morning and evening) for 10 days.

The study's primary objective is to evaluate whether the intensified omeprazole treatment reduces the average daily ileostomy fluid output in the first three days after surgery. Additional objectives include assessing how quickly stoma output stabilizes (defined as output less than 1400 ml/day for three consecutive days), comparing the incidence of dehydration-related complications such as electrolyte imbalances, evaluating differences in hospital stay duration, and monitoring the rates of rehospitalization within 30 days after discharge.

Participants in both groups will undergo daily monitoring of their ileostomy output and regular blood tests to check electrolyte levels during their hospital stay. After discharge, participants will continue to be followed for 30 days through outpatient visits or telephone consultations to monitor any further complications or health issues.

The findings of this study could provide crucial evidence regarding the benefits of intensified omeprazole therapy. If proven effective, this approach may significantly improve patient outcomes, reduce the frequency of complications associated with high-output stomas, shorten hospital stays, and lower healthcare costs related to postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled for elective or emergency surgery requiring end or loop ileostomy formation
* Able and willing to provide written informed consent
* No contraindications to omeprazole use

Exclusion Criteria:

* Pregnancy or lactation
* Known hypersensitivity or allergy to proton pump inhibitors (including omeprazole)
* Conditions preventing accurate measurement of daily ileostomy output

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
difference in mean ileostomy output (ml/24h) between postoperative days (POD) 1-3 between the experimental and control groups | from stoma creation to postoperative day 3
  The primary endpoint is the difference in mean ileostomy output (ml/24h) between postoperative days (POD) 1-3 between the experimental and control groups, after excluding patients with minimal output (<200 ml in any POD 1-3). A clinically significant reduction in output is defined as ≥250 ml/day.

SECONDARY OUTCOMES:
Proportion of patients meeting the criteria for high-output stoma | 1 month from stoma creation
  Proportion of patients meeting the criteria for high-output stoma (HOS ≥1400 ml/day) on consecutive postoperative days.
Time to stabilization of ileostomy output | 1 month from stoma creation
  Time to stabilization of ileostomy output (defined as output consistently <1400 ml/day for three consecutive days).
Incidence of dehydration-related complications | 30 days post discharge after stoma creation
  Incidence of dehydration-related complications (hyponatremia, hypokalemia). Hyponatremia will be evaluated by the number of hyponatremia incidents during the hospitalization and 30 days after discharge. Hypokalemia will be evaluated by the total sum of supplementation (g) needed and the number of hypokalemia incidents during the hspitalization.
Total length of hospitalization | 30 days post discharge after stoma creation
  Length of initial hospital stay (LOS - length of stay), rehospitalization rate within 30 days post-discharge, and total length of hospitalization (TLOS - total length of stay).

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław Kobiela, Professor, Study Chair — MUG Division of General Surgery
Locations (2):
- Poland (2):
  - Department of Oncological, Transplant and General Surgery, Univeristy Clinical Center, Gdansk, Pomeranian Voivodeship
  - Clinical Department of Oncologic Surgery with a Subdivision of Breast, Skin, and Soft Tissue Tumor Surgery PCK Maritime Hospital, Gdynia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeppesen PB, Staun M, Tjellesen L, Mortensen PB. Effect of intravenous ranitidine and omeprazole on intestinal absorption of water, sodium, and macronutrients in patients with intestinal resection. Gut. 1998 Dec;43(6):763-9. doi: 10.1136/gut.43.6.763. PMID 9824602
- [Background] Fujino S, Miyoshi N, Ohue M, Takahashi Y, Yasui M, Sugimura K, Akita H, Takahashi H, Kobayashi S, Yano M, Sakon M. Prediction model and treatment of high-output ileostomy in colorectal cancer surgery. Mol Clin Oncol. 2017 Sep;7(3):468-472. doi: 10.3892/mco.2017.1336. Epub 2017 Jul 19. PMID 28894582
- [Background] Lederhuber H, Massey LH, Kantola VE, Siddiqui MRS, Sayers AE, McDermott FD, Daniels IR, Smart NJ. Clinical management of high-output stoma: a systematic literature review and meta-analysis. Tech Coloproctol. 2023 Dec;27(12):1139-1154. doi: 10.1007/s10151-023-02830-1. Epub 2023 Jun 18. PMID 37330988
- [Background] Nightingale J, Woodward JM; Small Bowel and Nutrition Committee of the British Society of Gastroenterology. Guidelines for management of patients with a short bowel. Gut. 2006 Aug;55 Suppl 4(Suppl 4):iv1-12. doi: 10.1136/gut.2006.091108. No abstract available. PMID 16837533